CLINICAL TRIAL: NCT03587389
Title: An Open Single-arm Interventional Study to Identify the Influence of Human Genetic Variation on Early Transcriptional Responses and Protective Immunity Following Immunization With Rotarix Rotavirus Vaccine in Infants in HCM City in Vietnam
Brief Title: Response to Rotavirus Vaccine in Infants in Ho Chi Minh City in Vietnam
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Hung Vuong Hospital (Other); Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other); Children's Hospital Number 1, Ho Chi Minh City, Vietnam (Other); Wellcome Sanger Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21EN
Record Dates: First submitted 2018-04-17; First posted 2018-07-16 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Rotavirus; Diarrhea
Keywords: Rotavirus; Vaccine; Diarrhea; Host genetics
MeSH Terms: conditions — Diarrhea | interventions — RIX4414 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rotavirus vaccine (Experimental): The Rotarix vaccine package consist of 1.5 ml of oral suspension in a pre-filled oral applicator (type I glass) with a plunger stopper (rubber butyl) and a protective tip cap (rubber butyl) in pack sizes of 1.
  The vaccination course consists of two doses. The first dose may be administered from the age of 6 weeks. There should be an interval of at least 4 weeks between doses. The vaccination course should preferably be given before 16 weeks of age, but must be completed by the age of 24 weeks. Rotarix is for oral use only and should under no circumstancies be injected.
  All participating infants will receive two doses of Rotarix vaccine following the standard Rotarix immunization protocol.
  Interventions: Biological: Rotarix vaccine

INTERVENTIONS:
Biological: Rotarix vaccine — In this study, the 1st dose of Rotarix vaccine will be administered when infants are at ages between weeks 8-9 and the 2nd dose is 28-37 days after the 1st dose, which means that there is an interval of 28-37 days or 4-5 weeks between doses. A reminding call will be set at about 4 weeks after the 1st dose to remind parents to bring their children back to Hung Vuong Hospital for the 2nd dose of Rotarix to ensure the completion of the 2nd dose of Rotarix vaccine.

SUMMARY:
The primary objective is to measure the effect of host human genetics on the resulting immunological responses and long-term protection following rotavirus immunization of a study population of infants in Ho Chi Minh City, Vietnam.

The secondary objectives are to assess the temporal immunological responses following rotavirus vaccination, and to investigate the role of maternally derived antibodies, and other factors that could potentially affect immunological responses following rotavirus vaccination. Also to assess infecting rotavirus genotypes in the vaccine failure cases.

DETAILED DESCRIPTION:
This study will be an open single arm, single centre, interventional study conducted in Ho Chi Minh City, Vietnam. A sample size of 1,000 infants will be recruited to the study between 8 to 9 weeks (which is around 2 months) of age. These infants will receive two doses of the rotavirus vaccine, Rotarix with an interval of 28-37 days (or 4-5 weeks). The parents will be requested to bring the infants 2-3 days following each Rotarix vaccination to receive the standard EPI vaccinations. The infants will then be under passive and active surveillance for rotavirus-associated diarrhoea until 18 months of age. Blood samplings during pre and post vaccination and at 6, 12 and 18 month old visits will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Infants (both males and females) between 8 and 9 weeks (i.e. approximately 2 months) of age who are attending Hung Vuong Hospital to receive their standard EPI vaccinations.
* Currently registered residents of Districts 5 (where Hung Vuong Hospital is located) or 1, 6, 8, 10, or 11 (districts that are neighbouring district 5) in Ho Chi Minh city, with no specific intention of relocating in the next 12 months.
* Informed consent to be enrolled in the study and comply with study procedures, including host genetic studies.

Exclusion Criteria:

* Refusal of consent.
* Parent/ guardian under the age of 18.
* Premature (i.e. gestation period <37 weeks).
* Infants who have already been immunized with either a rotavirus vaccine or the standard 2-month EPI vaccinations.
* History of hypersensitivity to any components of the vaccine or adverse vaccine event.
* History of intussusception or congenital malformation of the gastrointestinal tract in the child that is likely to predispose child to intussusception.
* History of severe combined immunodeficiency disease (SCID), acquired immune deficiency syndrome (AIDS) or Human immunodeficiency virus (HIV) positivity, or other known immunodeficiency syndromes that may place the child at risk during immunisation.

Ages: 8 Weeks to 9 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 818 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
The rotavirus vaccine failure events during the time period from recruitment to 18 months of age. | from the recruitment to 18 months of age after the first dose of vaccination
  The primary endpoint is to measure the proportion of rotavirus vaccine failure events during the time period from recruitment to 18 months of age after the first dose of vaccination.

SECONDARY OUTCOMES:
Quantification of the antibody response following immunization | data collected during 7 site visits (Visit 1: Rotarix Dose 1, Visit 2: 2-3 after Visit 1, Visit 3: 28-37 days after Visit 1, Visit 4: 2-3 days after Visit 3, Visit 5: 6 months old, Visit 6: 12 months old, Visit 7: 18 months old)
  The temporal kinetics of rotavirus-specific antibody responses following immunization will be measured using virus-binding enzyme-linked immunosorbent assay (ELISA), which will be used to investigate the effect of host genetics, maternally transferred antibodies, and geospatial and epidemiological factors on the humoral response following vaccination.
Assessment of infecting rotavirus genotypes in vaccine failure cases | from the recruitment to 18 months of age after the first dose of vaccination
  The rotavirus genotypes in vaccine failure cases will be assessed to investigate whether vaccine failure cases are a result of varying rotavirus genotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Baker, Professor, Principal Investigator — Oxford University Clinical Research Unit
Locations (1):
- Hung Vuong Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided